CLINICAL TRIAL: NCT03569436
Title: Efficacy and Safety of Nivolumab in Recurrent or Metastatic Head and Neck Cancer (HNC) Patients - Japanese Real-world Data Through Clinical Chart Review
Brief Title: Effectiveness and Safety of Nivolumab in Participants That Have Head and Neck Cancer That Has Come Back or Has Spread
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-8DD
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Cancer of Head and Neck; Cancer of the Head; Cancer of the Neck
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic head and neck participants in Japan: Study in Japan targeting recurrent/metastatic HNC patients who are treated with nivolumab

SUMMARY:
Non-interventional study in Japan of participants with HNC recurring or that has spread and who are treated with nivolumab

ELIGIBILITY:
Inclusion Criteria:

* Recurrent/metastatic HNC patients with disease progression on or after a platinum-based therapy treated with nivolumab at least once from 01-Jul-2017 through 31-Dec-2017

Exclusion Criteria:

* History of participation in any clinical trials prior- or post-nivolumab treatment

Other protocol defined inclusion/exclusion criteria could apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Recurrent/Metastatic (R/M) squamous cell carcinoma of the head and neck (SCCHN) participants on nivolumab who progressed on or after platinum therapy
Sampling Method: Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Distribution of drug therapy treatment information | 6 months
Distribution of non-drug therapy treatment information | 6 months
Distribution of clinical laboratory testing | 6 months
Distribution of participant information | 6 months
Distribution of non-medication therapy treatment history | 12 months
Distribution of therapeutic history | 12 months
Overall survival | 12 months
Progression free survival | 12 months
Objective response rate | 12 months
Duration of response | 12 months

SECONDARY OUTCOMES:
Incidence of AE's | Up to 12 months
Incidence of serious AE's | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Tokyo, Japan

REFERENCES:
- [Derived] Kariya S, Shimizu Y, Hanai N, Yasumatsu R, Yokota T, Fujii T, Tsukahara K, Yoshida M, Hanyu K, Ueda T, Hirakawa H, Takahashi S, Ono T, Sano D, Yamauchi M, Watanabe A, Omori K, Yamazaki T, Monden N, Kudo N, Arai M, Yonekura S, Asakage T, Fujiwara A, Yamada T, Homma A. Effectiveness of nivolumab affected by prior cetuximab use and neck dissection in Japanese patients with recurrent or metastatic head and neck cancer: results from a retrospective observational study in a real-world setting. Int J Clin Oncol. 2021 Jun;26(6):1049-1056. doi: 10.1007/s10147-021-01900-4. Epub 2021 Apr 8. PMID 33830342
- [Derived] Hanai N, Shimizu Y, Kariya S, Yasumatsu R, Yokota T, Fujii T, Tsukahara K, Yoshida M, Hanyu K, Ueda T, Hirakawa H, Takahashi S, Ono T, Sano D, Yamauchi M, Watanabe A, Omori K, Yamazaki T, Monden N, Kudo N, Arai M, Sakurai D, Asakage T, Doi I, Yamada T, Homma A. Effectiveness and safety of nivolumab in patients with head and neck cancer in Japanese real-world clinical practice: a multicenter retrospective clinical study. Int J Clin Oncol. 2021 Mar;26(3):494-506. doi: 10.1007/s10147-020-01829-0. Epub 2020 Nov 21. PMID 33219460
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm